CLINICAL TRIAL: NCT05113433
Title: Effects of Different Time Period of Standing Frame on Spasticity and Gait in Children With Spastic Cerebral Palsy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shifa Tameer-e-Millat University (Other)
Responsible Party: Principal Investigator, Nouman Khan, Lecturer, Shifa Tameer-e-Millat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Anum Shahzadi 159-21
Record Dates: First submitted 2021-11-02; First posted 2021-11-09 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Spastic Cerebral Palsy; Spastic Gait
Keywords: Cerebral Palsy; Modified Ashworth scale; 6 minute walk test
MeSH Terms: conditions — Cerebral Palsy; Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group a (Experimental): 15 minute on standing frame .
  Interventions: Other: conventional physical therapy; Other: standing frame.
- group b (Experimental): 30 minute on standing frame .
  Interventions: Other: conventional physical therapy; Other: standing frame.
- group c (Experimental): 45 minute on standing frame.
  Interventions: Other: conventional physical therapy; Other: standing frame.
- group d (Experimental): 60 minute on standing frame.
  Interventions: Other: conventional physical therapy; Other: standing frame.

INTERVENTIONS:
Other: conventional physical therapy — muscle strengthening i.e. isometrics of lower limb muscles. 5 sets/rep and 2 sets/ session.
  stretching of lower limb muscles . 5sets/rep and 2 sets/session.
Other: standing frame. — muscle strengthening i.e. isometrics of lower limb muscles. 5 sets/rep and 2 sets/ session.
  stretching of lower limb muscles . 5sets/rep and 2 sets/session. sanding on standing frame for different time period according to group with upper limb activities lie box and blocks , cones and theraputty .

SUMMARY:
Cerebral palsy is a neurological disorder with abnormalities in muscle tone, movement disorders and motor incapability. It attributes to harm to the growing brain. Cerebral approach including brain and its palsy referred to weakness and problems while using the muscles. It is characterized by way of the incapability to normally control motor features, and it has. the capacity to have an impact on the general improvement of a child with the aid of affecting the child's capability to explore, talk, learn, and grow to be independent. Spastic CP is the most common type among children and debts for almost 77% among all instances. It is the major problem in CP child making movement difficult or even impossible.

DETAILED DESCRIPTION:
Cerebral palsy itself is not considered as a. progressive disease rather it is a medical. expression that may trade with time as the brain grows. It is attributed as the physical disability that is commonly present in children whose diagnosis can be made. before 6 months. Cerebral palsy is mostly considered as the commonplace physical incapacity among children .and it impacts almost 2 -2.5/1000 children born in United State of America. Population based information displays that the percentage of intense cases of CP is very high among low and middle earned international countries. Children with CP born in low offerings .Children with cerebral palsy mostly have spastic syndrome in common. Prolong sustain stretch is an effective treatment traditionally used to reduce spasticity. We can use the effect of frame and gravity or automatically, the usage of device or splints to carry out sustain stretch manually. A standing frame is a mechanical (vintage) or mechatronic (new) equipment, that has as principal aim to accurate the incapacity of certain individual for assuming the body's vertical position.

The type of cerebral palsy relies upon on the kind of movement disorders in children affecting the body parts. The classification of CP which is topographically involves:

Quadriplegic Hemiplegic Diplegic Monoplegic And triplegic cerebral palsy Clinical history may help an early diagnosis which involves the use of neuroimaging, standardized tests with neurological and motor aspects which indicates congruent ordinary findings indicating cerebral palsy. The importance of spark off referral need to be recognized by the clinicians to be specifically diagnostic before the start of intervention so that treatment can be optimized for the prevention of secondary complications. Types of CP contributes in the early diagnosis with presence of epilepsy, a larger degree of motor incapacity, and cerebral abnormalities in ultrasonography. There is no association between gestational and diagnostic age. Neuroimaging is presently endorsed as a general assessment. MRI showing excessive abnormality in white matter had a strong association with CP as compared to general movements present .MRI with respect to its diagnostic value is not as better as consecutive ultrasonography, the reason behind this fact is that MRI is much demanding, but MRI in daily routine is not going to turn out as a standard exercise.

ELIGIBILITY:
Inclusion Criteria:

* Spastic CP with age limit between 4-14 years.
* Both genders.
* At least 40° knee flexion.
* Sitting achieved on ground.
* mass at least with grade 3.

Exclusion Criteria:

* Children with knee flexor contractures > 60°.
* Hip flexor contractures > 60°.
* Planter flexor contractures > 30°.
* Severe mental retardation.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-11-02 (Estimated); Primary Completion 2021-12-02 (Estimated); Study Completion 2021-12-10 (Estimated)

PRIMARY OUTCOMES:
modified ashworth scale. | 4 weeks
  mas used to assess spasticity of lower limb muscles bilaterally i.e. hip flexors, hip extensors hip abductors hip adductors , ankle dorsiflexors and ankle planter flexiors.
6 minute walk test. | 4 weeks
  6 minute walk test to assess gait. walk for 6 minute . children can take rest but time will not be stopped. measure distance in meters.

CONTACTS AND LOCATIONS:
Overall Officials: Shafaq Altaf, Phd*, Principal Investigator — Shifa tameer e millat university Islamabad
Locations (1):
- Shifa tameer e millat university, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Audu O, Daly C. Standing activity intervention and motor function in a young child with cerebral palsy: A case report. Physiother Theory Pract. 2017 Feb;33(2):162-172. doi: 10.1080/09593985.2016.1265621. Epub 2017 Jan 10. PMID 28071965
- [Background] Bar-On L, Molenaers G, Aertbelien E, Van Campenhout A, Feys H, Nuttin B, Desloovere K. Spasticity and its contribution to hypertonia in cerebral palsy. Biomed Res Int. 2015;2015:317047. doi: 10.1155/2015/317047. Epub 2015 Jan 11. PMID 25649546
- [Background] Bearden DR, Monokwane B, Khurana E, Baier J, Baranov E, Westmoreland K, Mazhani L, Steenhoff AP. Pediatric Cerebral Palsy in Botswana: Etiology, Outcomes, and Comorbidities. Pediatr Neurol. 2016 Jun;59:23-9. doi: 10.1016/j.pediatrneurol.2016.03.002. Epub 2016 Mar 17. PMID 27114082
- [Background] Blackmore AM, Boettcher-Hunt E, Jordan M, Chan MD. A systematic review of the effects of casting on equinus in children with cerebral palsy: an evidence report of the AACPDM. Dev Med Child Neurol. 2007 Oct;49(10):781-90. doi: 10.1111/j.1469-8749.2007.00781.x. PMID 17880650
- [Background] Capati V, Covert SY, Paleg G. Stander Use for an Adolescent with Cerebral Palsy at GMFCS Level with Hip and Knee Contractures. Assist Technol. 2020 Nov 1;32(6):335-341. doi: 10.1080/10400435.2019.1579268. Epub 2019 Apr 4. PMID 30945990
- [Background] Caulton JM, Ward KA, Alsop CW, Dunn G, Adams JE, Mughal MZ. A randomised controlled trial of standing programme on bone mineral density in non-ambulant children with cerebral palsy. Arch Dis Child. 2004 Feb;89(2):131-5. doi: 10.1136/adc.2002.009316. PMID 14736627
- [Background] Dalembert G, Brosco JP. Do politics affect prevalence? An overview and the case of cerebral palsy. J Dev Behav Pediatr. 2013 Jun;34(5):369-74. doi: 10.1097/DBP.0b013e31829455d8. PMID 23751888
- [Background] Duke R, Eyong K, Burton K, MacLeod D, Dutton GN, Gilbert C, Bowman R. The effect of visual support strategies on the quality of life of children with cerebral palsy and cerebral visual impairment/perceptual visual dysfunction in Nigeria: study protocol for a randomized controlled trial. Trials. 2019 Jul 10;20(1):417. doi: 10.1186/s13063-019-3527-9. PMID 31291989
- [Background] Elnaggar RK, Elbanna MF, Mahmoud WS, Alqahtani BA. Plyometric exercises: subsequent changes of weight-bearing symmetry, muscle strength and walking performance in children with unilateral cerebral palsy. J Musculoskelet Neuronal Interact. 2019 Dec 1;19(4):507-515. PMID 31789302
- [Background] Franki I, Bar-On L, Molenaers G, Van Campenhout A, Craenen K, Desloovere K, Feys H, Pauwels P, De Cat J, Ortibus E. Tone Reduction and Physical Therapy: Strengthening Partners in Treatment of Children with Spastic Cerebral Palsy. Neuropediatrics. 2020 Apr;51(2):89-104. doi: 10.1055/s-0039-3400987. Epub 2019 Nov 27. PMID 31777043
- [Background] Goodwin J, Lecouturier J, Basu A, Colver A, Crombie S, Smith J, Howel D, McColl E, Parr JR, Kolehmainen N, Roberts A, Miller K, Cadwgan J. Standing frames for children with cerebral palsy: a mixed-methods feasibility study. Health Technol Assess. 2018 Sep;22(50):1-232. doi: 10.3310/hta22500. PMID 30234480